CLINICAL TRIAL: NCT04748068
Title: Use of Glidesheath Slender to Reduce Radial Artery Occlusion Following 7 French Transradial Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7F Glidesheath Slender
Record Dates: First submitted 2021-01-25; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Radial Artery Occlusion; Coronary Artery Disease
Keywords: Radial artery occlusion; 7-Fr radial sheath; Transradial Coronary Intervention
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glidesheath Slender (Experimental): The transradial procedure will be performed using the 7-Fr glidesheath slender (studied sheath)
  Interventions: Device: 7-Fr Glidesheath Slender
- Standard sheath (Active Comparator): The transradial procedure will be performed using the standard 7- French radial sheath (comparator sheath)
  Interventions: Device: Cordis 7-Fr radial sheath

INTERVENTIONS:
Device: 7-Fr Glidesheath Slender — The 7 Fr Glidesheath Slender is a recently developed thin-walled radial sheath. It combines an ID of 2.46 mm, with an OD of 2.79 mm, representing thereby the thinnest 7 Fr sheath currently available on the market
  Other Names: Glidesheath Slender, Terumo, Tokyo, Japan
  Arms: Glidesheath Slender
Device: Cordis 7-Fr radial sheath — Avanti+ Catheter Sheath Introducer, Cordis, USA, outer diameter: 3.02 mm
  Arms: Standard sheath

SUMMARY:
The objective of this study is to determine the rate of early radial artery occlusion following 7-French(7-Fr) transradial coronary intervention using a new Terumo (Tokyo, Japan) Glidesheath Slender, in comparison with the currently used 7-Fr radial sheath.

DETAILED DESCRIPTION:
Based on previously reported studies the rates of radial artery occlusion using a standard 7-Fr sheath is around 12%, compared to the previous studies of the Glidesheath Slender (see reference in the citations), the rate of radial artery occlusion was reported less than 5%. To prove Slender sheaths are superior to traditional ones, the sample size was estimated according to this, the class I error (α) is set as 0.05 on both sides, and the test efficiency (β) is set as 80%, then at least 248 patients are needed in each group.

This study will be a prospective randomized, single-blinded (patient-blinded) study, comparing the rate of radial artery occlusion between the 7-Fr Glidesheath Slender (Terumo, Japan) and the standard 7-Fr radial sheath (cordis, USA) in patients undergoing complex transradial coronary intervention.

The study will enroll patients who will undergo elective complex percutaneous coronary intervention (PCI) via 7-Fr transradial approach at Fuwai Hospital National Center for Cardiovascular Diseases.

A baseline clinical vascular & ultrasound assessment will be performed prior to the procedure to document patency of the radial artery.

Patients will be randomized in 1:1 fashion to either receive the 7-Fr Terumo Glidesheath Slender versus the currently used 7-Fr sheath.

The standard angiogram/ PCI will be performed as per usual practice. Following the PCI, clinical vascular assessment as well as an ultrasound will be performed prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary PCI via 7-Fr transradial approach
* Informed consent
* the patency of radial artery confirmed by ultrasound

Exclusion Criteria:

* The abnormal of radial artery confirmed by ultrasound
* Previous failed radial access.
* Known bleeding disorder or hypercoagulable condition
* Cardiogenic shock

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Radial artery occlusion | 24 hours
  Evaluated clinically and by ultrasound

SECONDARY OUTCOMES:
Vascular access site complications | 24 hours
  Includes: bleeding or hematoma, pseudoaneurysm, artery dissection, arteriovenous fistula, compartment syndrome of the forearm
Radial artery spasm | 24 hours
  Radial artery spasm
Procedure success | 24 hours
  completion of the planned procedure through the initially selected radial access route
The degree of pain at the puncture site | 24 hours
  Scored on a scale of 1-10 scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Kefei Dou, MD,PhD, Principal Investigator — Fuwai Hospital National Center for Cardiovascular Diseases; Chenggang Zhu, MD,PhD, Principal Investigator — Fuwai Hospital National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rashid M, Kwok CS, Pancholy S, Chugh S, Kedev SA, Bernat I, Ratib K, Large A, Fraser D, Nolan J, Mamas MA. Radial Artery Occlusion After Transradial Interventions: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Jan 25;5(1):e002686. doi: 10.1161/JAHA.115.002686. PMID 26811162
- [Background] Bernat I, Aminian A, Pancholy S, Mamas M, Gaudino M, Nolan J, Gilchrist IC, Saito S, Hahalis GN, Ziakas A, Louvard Y, Montalescot G, Sgueglia GA, van Leeuwen MAH, Babunashvili AM, Valgimigli M, Rao SV, Bertrand OF; RAO International Group. Best Practices for the Prevention of Radial Artery Occlusion After Transradial Diagnostic Angiography and Intervention: An International Consensus Paper. JACC Cardiovasc Interv. 2019 Nov 25;12(22):2235-2246. doi: 10.1016/j.jcin.2019.07.043. PMID 31753298
- [Background] Aminian A, Iglesias JF, Van Mieghem C, Zuffi A, Ferrara A, Manih R, Dolatabadi D, Lalmand J, Saito S. First prospective multicenter experience with the 7 French Glidesheath slender for complex transradial coronary interventions. Catheter Cardiovasc Interv. 2017 May;89(6):1014-1020. doi: 10.1002/ccd.26773. Epub 2016 Aug 27. PMID 27567021
- [Background] Isawa T, Horie K, Honda T, Taguri M, Tada N. Slender Sheath/Guiding Catheter Combination vs. Sheathless Guiding Catheter for Acute Coronary Syndrome: A Propensity-Matched Analysis of the Two Devices. J Interv Cardiol. 2020 Aug 14;2020:8216831. doi: 10.1155/2020/8216831. eCollection 2020. PMID 32863791
- [Background] Saito S, Ikei H, Hosokawa G, Tanaka S. Influence of the ratio between radial artery inner diameter and sheath outer diameter on radial artery flow after transradial coronary intervention. Catheter Cardiovasc Interv. 1999 Feb;46(2):173-8. doi: 10.1002/(SICI)1522-726X(199902)46:23.0.CO;2-4. PMID 10348538
- [Background] Costa F, van Leeuwen MA, Daemen J, Diletti R, Kauer F, van Geuns RJ, Ligthart J, Witberg K, Zijlstra F, Valgimigli M, Van Mieghem NM. The Rotterdam Radial Access Research: Ultrasound-Based Radial Artery Evaluation for Diagnostic and Therapeutic Coronary Procedures. Circ Cardiovasc Interv. 2016 Feb;9(2):e003129. doi: 10.1161/CIRCINTERVENTIONS.115.003129. PMID 26839392
- [Derived] Wang H, Wang HY, Wu SY, Yin D, Feng L, Song WH, Wang HJ, Zhu CG, Dou KF. Effect of Thin-Walled Radial Sheath for Large-Bore Access On Reducing Periprocedural Radial Artery Occlusion Following Complex PCI: The REDUCE-RAO Randomized Trial. Rev Cardiovasc Med. 2022 Sep 28;23(10):329. doi: 10.31083/j.rcm2310329. eCollection 2022 Oct. PMID 39077135